CLINICAL TRIAL: NCT03100396
Title: Direct Reporting of Awareness in Maternity Patients: a Prospective Evaluation of Accidental Awareness Under General Anaesthesia in Obstetric Surgery Patients
Brief Title: Direct REporting of Awareness in MaternitY Patients
Acronym: DREAMY
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: St George's, University of London (Other)
Responsible Party: Sponsor
Other Study IDs: 16.0063; 203113 (Other: IRAS ID)
Record Dates: First submitted 2017-03-07; First posted 2017-04-04 (Actual); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Awareness, Anesthesia; Obstetric Anesthesia Problems
MeSH Terms: conditions — Intraoperative Awareness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
DREAMY is a prospective, multi-centre observational cohort study using a mixed methods approach to provide quantitative and qualitative data on accidental awareness under general anaesthesia (AAGA) in obstetric surgery patients. Obstetric patients undergoing surgery, such as emergency caesarian section under general anaesthesia, are thought to be at higher risk than any other surgical cohorts for AAGA. Patients recruited to the study will be screened for AAGA using a standardised questionnaire on three occasions over 30 days. Follow up with structured interviews for all AAGA patients will occur over 12 months.

DETAILED DESCRIPTION:
Background: The challenges of obstetric general anaesthesia practice - including the use of rapid sequence induction, neuromuscular blockade and short duration between anaesthetic induction and start of surgery - may contribute to a higher risk of awareness under general anaesthesia (AAGA) in these patients. The 2014 Royal College of Anaesthetists/Association of Anaesthetists of Great Britain and Ireland National Audit Project 5 highlighted a higher risk of spontaneously reported AAGA in obstetric patients, but it remains unclear what the full (i.e. non-spontaneously reported) risk is. The aim of DREAMY is to establish the incidence of AAGA following general anaesthesia in obstetric surgery patients.

Methods: A standardised Brice questionnaire will be used to screen for recall of intraoperative events in women meeting the eligibility requirements. Questions asked are:

1. What is the last thing you remember before going to sleep?
2. What is the first thing you remember after waking up?
3. Do you remember anything between going to sleep and waking up?
4. Did you dream during your procedure?
5. What was the worst thing about your operation?

The validity of the AAGA incidence will be improved by repetition of the questionnaire on three occasions over thirty days and triangulating using structured follow up interviews in all participants reporting AAGA in questionnaire responses. Participants will be followed up over 12 months and asked for self-reported symptoms of post-traumatic stress disorder (PTSD) using the PCL-5 checklist. The research is being run as a multi-centre, descriptive study over 12 months. General condition and details of the anaesthetic procedure will also be recorded for a logistic regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* Female adults (≥18 years) of ≥ 24/40 gestation
* Receiving general anaesthesia (de novo or regional anaesthesia converted to GA) for surgery with an obstetric indication (e.g. emergency caesarean section, manual removal of placenta, examination under anaesthesia)

Exclusion Criteria:

* Patients too unwell or confused to be able to complete the questionnaire
* Patient refusal
* General anaesthesia for non-obstetric indication (e.g. colorectal or orthopaedic surgery in a pregnant patient)
* Surgery ≥48 hours post-partum
* Unable to communicate verbally/in writing in English language

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Study Population: Women undergoing obstetric-indication surgery under general anaesthesia
Sampling Method: Non-Probability Sample
Enrollment: 3100 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2019-08-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of accidental awareness under general anaesthesia | 30 days
  Unintended awareness under general anaesthesia being reported following direct questioning with a Brice questionnaire

SECONDARY OUTCOMES:
Incidence and types of dreams under anaesthesia | 30 days
  Qualitative data on each awareness event; including recall, timing, understanding and emotional response
Incidence of post-traumatic stress disorder (PCL-5 checklist) | 12 months
  Incidence of post-traumatic stress disorder symptoms following awareness events
Predictors of post-traumatic stress disorder based on patient characteristics and type of awareness event | 12 months
  Characteristics associated with post-traumatic stress disorder following anaesthesia with awareness and without awareness
Predictors of awareness based on patient, surgical and anaesthetic characteristics | 12 months
  Modifiable and non-modifiable characteristics associated with awareness
Comparison of direct questioning vs. semi-structured interview schedule approaches to assessing the incidence of awareness | 12 months
  Response from the Brice questionnaire will be assessed against responses gathered in during semi-structured interview schedules

CONTACTS AND LOCATIONS:
Overall Officials: Peter M Odor, Study Chair — St George's, University of London
Locations (1):
- St. George's University Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Odor PM, Bampoe S, Lucas DN, Moonesinghe SR, Andrade J, Pandit JJ; DREAMY Investigators Group. Protocol for direct reporting of awareness in maternity patients (DREAMY): a prospective, multicentre cohort study of accidental awareness during general anaesthesia. Int J Obstet Anesth. 2020 May;42:47-56. doi: 10.1016/j.ijoa.2020.02.004. Epub 2020 Feb 14. PMID 32139144